CLINICAL TRIAL: NCT03937323
Title: Immun Parameters and Flow Cytometry at Pancreatitis Patients
Brief Title: Immun Status at Pancreatitis Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Principal Investigator, Istanbul Training and Research Hospital
Other Study IDs: Pancreatitis immun status
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2020-07

CONDITIONS: Pancreatitis; Immune Suppression
Keywords: Pancreatitis; Lymphocyte subtypes; Cytokine
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Pancreatitis group: Patients with biliary pancreatitis
  Interventions: Other: Blood lymphocyte subtypes and serum cytokines
- Group 2: Control group,: Healthy volunteers
  Interventions: Other: Blood lymphocyte subtypes and serum cytokines

INTERVENTIONS:
Other: Blood lymphocyte subtypes and serum cytokines — Blood samples will be taken from the patients with biliary pancreatitis and healthy volunteers to perform flow-cytometric analysis and to determine the proinflammatory cytokines

SUMMARY:
Pancreatitis is a common complication especially in patients with gallbladder stones, most patients with biliary pancreatitis may recover spontaneously without sequelae, but in 10-20% of patients, the disease is severe and mortality rates of up to 30% are detected in these patients. In the evaluation of acute biliary pancreatitis, many scoring systems have been established (Atlanta, Ranson, APACHE, BISAP etc.) from past to present to determine morbidity and mortality of the disease.

In this study, the investigators aimed to evaluate the correlation between morbidity and mortality of acute biliary pancreatitis and serum proinflammatory cytokines with ELISA and lymphocyte subtypes with Flow-cytometry.

DETAILED DESCRIPTION:
Pancreatitis is a common complication especially in patients with gallbladder stones, most patients with biliary pancreatitis may recover spontaneously without sequelae, but in 10-20% of patients, the disease is severe and mortality rates of up to 30% are detected in these patients. In patients with severe pancreatitis, aggressive fluid replacement, organ damage follow-up, appropriate antibiotherapy, and endoscopic sphincterotomy and radiological interventions may be of great benefit. In the evaluation of acute biliary pancreatitis, many scoring systems have been established (Atlanta, Ranson, APACHE, BISAP etc.) from past to present to determine morbidity and mortality of the disease. There are limited number of studies in the literature about the immune parameters in the evaluation of acute pancreatitis. In a studies, serum inflammatory markers such as IL-1, IL-6 and CD4, CD8 T lymphocyte and Treg population were evaluated. It was reported that inflammatory markers, especially anti-inflammatory IL-10 levels were elevated in patients with acute pancreatitis, and CRP and IL-1β levels of inflammatory markers were higher in patients with organ failure. Treg cells are reported to be an independent prognostic factor in determining the severity of acute pancreatitis. There is only one study with a limited number of patients in whom PD-1 values in T lymphocytes and PD-L1 values in monocytes were determined in the literature. In this study, it is stated that PD-L1 can be used as a new marker in determining infectious complications. In patients diagnosed with acute biliary pancreatitis, determination of the course of the disease at the time of diagnosis is extremely important for treatment and survival.

In this study, the investigators aimed to evaluate the correlation between morbidity and mortality of acute biliary pancreatitis and serum proinflammatory cytokines with ELISA and lymphocyte subtypes with Flow-cytometry.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Diagnosis of acute biliary pancreatitis
* Sign the voluntary consent form

Exclusion Criteria:

* Being under 18 or older than 80
* Not signing the voluntary consent form
* Pancreatitis resulting from an interventional procedure (ERCP, surgery, etc.)
* Pregnant women
* Being a history of immunodeficiency
* Cancer history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with biliary pancreatitis will be classified into three subgroups according to Apache classification and also Healthy Volunteers will be control group.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Lymphocyte and monocyte subtypes | 1 day
  To determine T lymphocyte subtypes with Flow-Cytometry; T helper (CD4) (%) T cytotoxic (CD8) (%) NK cells (%) Classical monocytes Intermediate monocytes Non- Classical Monocytes
PD1,PDL1 | 1 day
  To determine percent of PD1 and PDL1 on T lymphocytes and monocytes with Flow-Cytometry

SECONDARY OUTCOMES:
Cytokines | 1 day
  To determineof IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1, IL-6, IL -8, IL-10, IL-12p (p70), IL-17A, IL-18, IL-,23 and IL-33 values with Flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc. Prof, Principal Investigator — Istanbul Training and Research Hospital
Locations (4):
- Turkey (Türkiye) (4):
  - Istanbul Traininng and Research Hospital, Istanbul
  - Hisar Hospital Intercontinental, Istanbul
  - Sisli Hamidiye Etfal Training and Research Hospital, Istanbul
  - Yeditepe University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
If the editors want to see our data we can share

REFERENCES:
- [Background] Wang W, Xiang HP, Wang HP, Zhu LX, Geng XP. CD4 + CD25 + CD127 high cells as a negative predictor of multiple organ failure in acute pancreatitis. World J Emerg Surg. 2017 Feb 2;12:7. doi: 10.1186/s13017-017-0116-7. eCollection 2017. PMID 28174597
- [Background] Yang Z, Zhang Y, Dong L, Yang C, Gou S, Yin T, Wu H, Wang C. The Reduction of Peripheral Blood CD4+ T Cell Indicates Persistent Organ Failure in Acute Pancreatitis. PLoS One. 2015 May 4;10(5):e0125529. doi: 10.1371/journal.pone.0125529. eCollection 2015. PMID 25938229
- [Background] Li J, Yang WJ, Huang LM, Tang CW. Immunomodulatory therapies for acute pancreatitis. World J Gastroenterol. 2014 Dec 7;20(45):16935-47. doi: 10.3748/wjg.v20.i45.16935. PMID 25493006